CLINICAL TRIAL: NCT05238506
Title: The Effect of Intravenous Lidocaine Infusion on Hemodynamic Reaction to Tracheal Intubation, as Well as Metabolic and Hormonal Response to Laparoscopic Procedure in Children: a Randomized Controlled Trial
Brief Title: Lidocaine VS Hemodynamic, Metabolic and Hormonal Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Maciej Kaszyński, physician, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Lido02
Record Dates: First submitted 2022-01-21; First posted 2022-02-14 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hemodynamic Response; Acute Appendicitis; Complication of Treatment; Opioid Consumption; Pneumoperitoneum
Keywords: multimodal analgesia; lidocaine; intravenous lidocaine; laparoscopic appendectomy; children; pediatric population; adjuvant; metabolic stress response; hormonal response
MeSH Terms: conditions — Appendicitis; Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The drug or placebo(normal saline) will be placed in a syringe by the principal investigator. Only principal investigator will be aware of the participants allocation. The principal investigator will not be involved in the process of: recruitment, providing an intervention, or outcomes assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Experimental): 1% lidocaine intravenous bolus of 0.15 ml/kg over 5 min before induction of anesthesia followed by lidocaine infusion at 0.15 ml/kg/h intraoperatively will be administered. The infusion will be discontinued before the patients' transfer to the postanesthesia care unit.
  Interventions: Drug: Intravenous lidocaine
- Control (Placebo Comparator): 0.9% NaCl intravenous bolus of 0.15 ml/kg over 5 min before induction of anesthesia followed by 0.9% NaCl infusion at 0.15 ml/kg/h intraoperatively will be administered. The infusion will be discontinued before the patients' transfer to the postanesthesia care unit.
  Interventions: Drug: Normal saline infusion

INTERVENTIONS:
Drug: Intravenous lidocaine — Intraoperative intravenous lidocaine infusion.
  Other Names: IVL
  Arms: Lidocaine
Drug: Normal saline infusion — Intraoperative intravenous normal saline infusion.
  Other Names: Placebo
  Arms: Control

SUMMARY:
Intravenous lidocaine - a potent local anesthetic with analgesic and anti- inflammatory properties has been shown to be an effective adjunct that reduces intra and postoperative opioid consumption and facilitates pain management in adults. In children population promising but limited evidence is available. The study has been planned to evaluate the efficacy of continuous intravenous infusion of lidocaine in alleviation of hemodynamic reaction to tracheal intubation, as well as metabolic and hormonal response to laparoscopic procedure in children.

DETAILED DESCRIPTION:
Laryngoscopy and endotracheal intubation are associated with noxious stimulation. Exacerbated circulatory system response may present as hypertension or arrhythmias including cardiac arrest. A sudden change in hemodynamic status connected with painful stimulation may precipitate deterioration in cerebral blood flow, especially in patients with intracranial hypertension (traumatic brain injury, intracranial hemorrhage, active hydrocephalus, etc). Many interventions have been applied to attenuate harmful hemodynamic reaction. One of them is intravenous lidocaine infusion. According to available data lidocaine is superior to placebo in attenuating systolic, diastolic and mean arterial pressure changes in children. Our study will focus on assessing hemodynamic stability preserving properties during induction of anesthesia and tracheal intubation. Blood pressure will be recorded and analyzed. The secondary aim is to examine intravenous lidocaine infusion in terms of reducing systemic response to surgical stress. Cortisol and glucose levels will be measured before skin incision, and immediately after the end of surgery. Side effects and serum lidocaine levels will be recorded to determine safety of the examined intervention. Similar pattern of infusion was investigated in RCT concerning children population - the toxic plasma level of 5 mcg/ml was not reached. Studies on children population have promising results but high quality randomized controlled trials are still missing. The proposed study has been planned to evaluate the efficacy of continuous infusion of lidocaine as an adjunct to standard general anesthesia (involving intravenous induction and opioid with sevoflurane maintenance) in attenuating hemodynamic reaction to tracheal intubation, as well as metabolic and hormonal response to surgical procedure in children undergoing laparoscopic appendectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class 1E, 2E, 3E;
* Patients undergoing laparoscopic appendectomy.

Exclusion Criteria:

* Allergy to local anesthetics or contraindications for the use of lidocaine;
* ASA physical status class 4E or higher;
* Severe cardiovascular disease;
* Preoperative bradycardia;
* Preoperative atrioventricular block;
* Renal failure;
* Chronic treatment with analgesics;
* Legal guardians' refusal.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Hemodynamic reaction to tracheal intubation | Before intubation - immediately after intubation.
  A change in arterial blood pressure more than 20% from baseline. The fractions of patients in each group will be compared.

SECONDARY OUTCOMES:
Metabolic response to laparoscopic procedure | First blood sample will be taken 5 minutes after tracheal intubation. Second blood sample will be taken just before extubation.
  Glucose [mg/dl] levels will be measured and compared before and after laparoscopic procedure.
Lidocaine blood level | First blood sample will be taken 5 minutes after tracheal intubation. Second blood sample will be taken just before extubation.
  Lidocaine level [mcg/ml] will be measured after initial bolus and just before the end of its infusion.
Side effects of lidocaine | From the beginning of drug infusion until transfer to the postanesthesia care unit (10 minutes after extubation).
  Side effects of lidocaine will be assessed by recording the rates of the following complications: arrythmia, hypotension (defined as <70th percentile for age), allergic reaction.
Hormonal response to laparoscopic procedure | First blood sample will be taken 5 minutes after tracheal intubation. Second blood sample will be taken just before extubation.
  Cortisol levels [mcg/dl] will be measured and compared before and after laparoscopic procedure.

OTHER OUTCOMES:
The requirement for opioids during anesthesia | From the induction of anesthesia through to postanesthesia care unit admission (10 minutes after extubation).
  Total amount of fentanyl in micrograms per kilogram body weight used during anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Kaszyński, Principal Investigator — Medical University of Warsaw
Locations (1):
- University Clinic Centre of Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, CSR
Time Frame: The study protocol will be available to other researchers continuously after its publication.
  The CSR will be hopefully publicated after the study completion.
Access Criteria: The datasets used and/or analysed during the study will be available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Qi DY, Wang K, Zhang H, Du BX, Xu FY, Wang L, Zou Z, Shi XY. Efficacy of intravenous lidocaine versus placebo on attenuating cardiovascular response to laryngoscopy and tracheal intubation: a systematic review of randomized controlled trials. Minerva Anestesiol. 2013 Dec;79(12):1423-35. Epub 2013 Jul 9. PMID 23839320
- [Background] El-Deeb A, El-Morsy GZ, Ghanem AAA, Elsharkawy AA, Elmetwally AS. The effects of intravenous lidocaine infusion on hospital stay after major abdominal pediatric surgery. A randomized double-blinded study. Egypt J Anaesth. 2013;29(3):225-230, doi: 10.1016/j.egja.2013.02.005.
- [Background] Kaszynski M, Lewandowska D, Sawicki P, Wojcieszak P, Pagowska-Klimek I. Efficacy of intravenous lidocaine infusions for pain relief in children undergoing laparoscopic appendectomy: a randomized controlled trial. BMC Anesthesiol. 2021 Jan 5;21(1):2. doi: 10.1186/s12871-020-01218-0. PMID 33397287
- [Derived] Kaszynski M, Stankiewicz B, Kalicka A, Mikolap K, Olszanecka M, Rybka Z, Witt P, Darowski M, Pagowska-Klimek I. Comparison of Opioid Consumption During Paediatric Anaesthesia with and Without a Mandatory Protocol: A Retrospective Cohort Study. J Clin Med. 2025 Oct 22;14(21):7481. doi: 10.3390/jcm14217481. PMID 41226876
- [Derived] Kaszynski M, Kuczerowska A, Pietrzyk J, Sawicki P, Witt P, Stankiewicz B, Darowski M, Pagowska-Klimek I. Influence of intravenous lidocaine infusion on haemodynamic response to tracheal intubation and metabolic-hormonal responses during laparoscopic procedures in children: a randomised controlled trial. BMC Anesthesiol. 2025 Jan 10;25(1):23. doi: 10.1186/s12871-024-02885-z. PMID 39794723